CLINICAL TRIAL: NCT03151603
Title: Reducing Antibiotic Use for Uncomplicated Urinary Tract Infection in General Practice by Treatment With Uva Ursi (UU)- a Comparative Effectiveness Trial
Acronym: REGATTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Karsten Gavenis, Quality Assurance Staff Unit Clinical Trials, University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01579
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Urinary Tract Infections
Keywords: Uva Ursi; fosfomycin; uncomplicated urinary tract infection of women
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uva Ursi (Experimental): placebo to fosfomycin: 3 g granules orally 1x1 (day 0)
  and
  Uva Ursi: 105 mg (Arctuvan®) 3x2 tablets orally from day 0 for 5 days
  Interventions: Drug: Arctuvan; Drug: Placebo to Fosfomycin
- fosfomycin (Active Comparator): fosfomycin (Monuril®): 3 g granules orally 1x1 (day 0),
  and
  placebo to Uva Ursi: 3x2 tablets orally from day 0 for 5 days
  If the patient returns with persistent/recurrent symptoms, antibiotic therapy according to the sensitivity test.
  Interventions: Drug: Fosfomycin; Drug: Placebo to Arctuvan

INTERVENTIONS:
Drug: Arctuvan — application of a herbal drug
  Arms: Uva Ursi
Drug: Fosfomycin — application of an antibiotic drug
  Arms: fosfomycin
Drug: Placebo to Arctuvan — application of Placebo to Arctuvan
  Arms: fosfomycin
Drug: Placebo to Fosfomycin — application of Placebo to Fosfomycin
  Arms: Uva Ursi

SUMMARY:
It is well known that "over-treatment" of straightforward infections should be avoided as far as possible. Evidence-based data on non antibiotic treatment options for common conditions are therefore needed urgently. This randomised-controlled double blind trial examines whether initial herbal treatment with Uva Ursi, and antibiotic treatment only if symptoms persist, reduces antibiotic consumption in uncomplicated urinary tract infections (UTI) without a negative effect on symptom course and rate of recurrent UTIs. In total, 430 patients presenting with typical UTI symptoms will be included by their GPs and receive randomised either herbal treatment with uva ursi (antibiotics only if symptoms persist), or initial antibiotic treatment. Patients record symptom severity and drug intake in a diary and complete a final questionnaire after 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Women (18-75 years) with suspected UTI
* at least two symptoms of UTI (dysuria, urgency of micturition, frequency, lower abdominal pain)
* Written informed consent

Exclusion Criteria:

* signs of complicated UTI (e. g. temperature > 38°C, loin tenderness)
* conditions that may lead to complicated infections (i.e. renal diseases, patients with urinary catheter)
* pregnancy/ breastfeeding
* current self-medication with UU preparations e.g. z.B. Cystinol®, Uvalysat®, Arctuvan®
* antibiotic use in the last 7 days
* previous UTI in the past 2 weeks
* history of pyelonephritis
* contraindications for trial drugs
* serious diseases
* inability to understand trial Information
* current participation in another clinical trial or participation in another clinical trial within the last 4 weeks

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
antibiotic courses | day 0-28
  number of antibiotic courses from day 0 to day 28
symptom burden | day 0-7
  symptom burden (AUC) from day 0 to day 7

SECONDARY OUTCOMES:
early relapses | day 0-14
  number of early relapses until day 14
recurrent UTI | day 15-28
  number of recurrent UTI day 15-28
symptom resolution | day 4 and 7
  number of patients with symptom resolution on day 4/7
symptom sum score by patients' questionnaire | day 0-7
  mean daily symptom sum scores from day 0 to day 7; Each of the symptoms dysuria, urgency, frequency and lower abdominal pain is scored daily on a five point scale from 0 "none" to 4 "very strong" in a patients' questionnaire.
symptom burden for dysuria | day 0-7
  symptom burden (AUC) for dysuria scored daily on a five point scale from 0 "none" to 4 "very strong", from day 0 to day 7
symptom burden positive urine culture | day 0-7
  symptom burden (AUC) day 0-7 of patients with positive urine culture
symptom burden negative urine culture | day 0-7
  symptom burden (AUC) day 0-7 of patients with negative urine culture
activity impairment by UTI symptoms, measured as AUC | day 0-7
  activity impairment by UTI symptoms (days 0-7), measured as AUC. Impairment by each UTI symptom is scored daily on a five point scale from 0 "none" to 4 "very strong".
painkillers | day 0-7
  use of painkillers (Defined Daily Dose (DDD) day 0-7)
patients taking painkillers | day 28
  number of patients taking painkillers
antibiotic use | day 0-28
  antibiotic use (defined daily dose (DDD) day 0-28)
UTI related visits | day 0-28
  number of UTI related visits day 0-28
UTI related sick leave | day 0-28
  number of days of UTI related sick leave day 0-28
patients with poor outcome: temperature | day 0-7
  number of patients with temperature >38°C, day 0-7, according to patients´ statement
patients with poor outcome: worsening symptoms | day 28
  number of patients with worsening symptoms (impairment in symptom score)
patients with poor outcome: prolonged symptoms | day 0-28
  number of patients with prolonged symptoms (> 7 days), day 0-28. Patients will be followed up until symptom resolution, defined as max. 1 score point on each symptom scale.
pyelonephritis | day 0-28
  number of pyelonephritis day 0-28, according to GP´s diagnosis
AE and SAE | day 0-28
  number of AE and SAE by system organ class day 0-28
patients with at least 1 AE/ 2 AE | day 28
  proportion of patients with at least 1 AE/ 2 AE
symptom burden for urgency | day 0-7
  symptom burden (AUC) for urgency scored daily on a five point scale from 0 "none" to 4 "very strong", from day 0 to day 7
symptom burden for frequency | day 0-7
  symptom burden (AUC) for frequency scored daily on a five point scale from 0 "none" to 4 "very strong", from day 0 to day 7
symptom burden for lower abdominal pain | day 0-7
  symptom burden (AUC) for lower abdominal pain scored daily on a five point scale from 0 "none" to 4 "very strong", from day 0 to day 7

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hummers-Pradier, Prof. Dr., Principal Investigator — University Medical Center Göttingen
Locations (47):
- Germany (47):
  - Hausarztpraxis Dr. Raby, Achim
  - General Practice Aden, Braunschweig
  - General Practice Scheffer, Braunschweig
  - General Practice Coutelle, Bremen
  - General Practice Schelp, Bremen
  - General Practice Dickow, Burgwedel
  - General Practice Kiwit-Putzer, Burgwedel
  - Praxis Zietz, Celle
  - General Practice Kutzsche, Emmerthal
  - Praxis Dr. Bahr, Gieboldehausen
  - General Practice Müller, Gillersheim
  - Institute of General Medicine, University Medical Center Goettingen, Göttingen
  - Praxisgemeinschaft Jacob / Kling, Göttingen
  - General Practice Keske, Göttingen
  - General Practice Koch, Göttingen
  - General Practice Kolb, Göttingen
  - General Practice Lang, Göttingen
  - General Practice Lückerath, Göttingen
  - Praxis Dr. Egner, Hanover
  - Institute of General Medicine, MHH Hannover, Hanover
  - General Practice Barth, Hanover
  - General Practice Löber, Hardegsen
  - Gemeinschaftspraxis Dres Schlesier / Eckhardt, Heilbad Heiligenstadt
  - Gemeinschaftspraxis Hartleb / Stöcking, Heilbad Heiligenstadt
  - Praxis Dr. Koch, Heilbad Heiligenstadt
  - Praxisgemeinschaft Seitz / Eckert, Herzberg
  - General Practice Wilde, Hildesheim
  - Praxisgemeinschaft Stoltz / Raddatz, Höxter
  - General Practice Beverungen, Höxter
  - Gemeinschaftspraxis Kasperczyk / Schindewolf-Lensch, Isernhagen-Süd
  - General Practice Franz, Katlenburg-Lindau
  - Praxis Dr. Ohlendorf, Langenhagen
  - General Practice Ertel, Langwedel
  - General Practice Wehrbein, Lemförde
  - General Practice Lindenblatt, Neustadt
  - Hausarztzentrum Nörten, Nörten-Hardenberg
  - General Practice Preiskorn, Rehburg-Loccum
  - General Practice Meier-Ahrens, Rosdorf
  - General Practice Woitschek, Salzgitter
  - General Practice Beulshausen, Sattenhausen
  - General Practice Schulte, Scheeßel
  - General Practice Böttcher, Schwanewede
  - General Practice Albrecht, Springe
  - General Practice Wolf, Uslar
  - General Practice Schmiemann, Verden an der Aller
  - General Practice Annweiler, Waake
  - General Practice Stegemann, Wunstorf

REFERENCES:
- [Derived] Gagyor I, Hummers E, Schmiemann G, Friede T, Pfeiffer S, Afshar K, Bleidorn J. Herbal treatment with uva ursi extract versus fosfomycin in women with uncomplicated urinary tract infection in primary care: a randomized controlled trial. Clin Microbiol Infect. 2021 Oct;27(10):1441-1447. doi: 10.1016/j.cmi.2021.05.032. Epub 2021 Jun 7. PMID 34111592
- [Derived] Afshar K, Fleischmann N, Schmiemann G, Bleidorn J, Hummers-Pradier E, Friede T, Wegscheider K, Moore M, Gagyor I. Reducing antibiotic use for uncomplicated urinary tract infection in general practice by treatment with uva-ursi (REGATTA) - a double-blind, randomized, controlled comparative effectiveness trial. BMC Complement Altern Med. 2018 Jul 3;18(1):203. doi: 10.1186/s12906-018-2266-x. PMID 29970072